CLINICAL TRIAL: NCT00329433
Title: The Use of Desirudin Versus Heparin for Thrombosis Prophylaxis in Cardiothoracic Surgery Patients
Brief Title: Study Comparing Desirudin With Heparin to Prevent Vein Clots After Heart and Lung Surgery
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Barnes-Jewish Hospital (Other); Canyon Pharmaceuticals, Inc. (Industry)
Responsible Party: Principal Investigator, Michael Avidan, Professor of Anesthesiology, Washington University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 05-0969
Record Dates: First submitted 2006-05-22; First posted 2006-05-24 (Estimated); Results first posted 2011-06-13 (Estimated); Last update posted 2019-03-05 (Actual); Status verified 2011-06

CONDITIONS: Deep Venous Thrombosis
Keywords: Deep venous thrombosis; DVT; Heparin induced thrombocytopenia; HIT; Direct thrombin inhibitor
MeSH Terms: conditions — Venous Thrombosis | interventions — desirudin; Heparin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Heparin (Active Comparator): Both groups of patients will receive study drug three times a day (TID) for DVT prophylaxis. The current TID schedule is 0900, 1300, and 2100. The patients who are randomized to the Heparin (standard of care) group will receive subcutaneous injections of heparin three times a day (0900, 1300 and 2100).
  Interventions: Drug: Heparin
- Desirudin (Iprivask™) (Experimental): Both groups of patients will receive study drug three times a day (TID) for DVT prophylaxis. The current TID schedule is 0900, 1300, and 2100. Patients who are randomized to the desirudin (study) group will receive 15 mg of subcutaneous desirudin twice a day (at 0900 and 2100). These patients will also receive an injection of normal saline placebo at 1300 so that patients in both groups will receive three injections at the same time points.
  Interventions: Drug: Desirudin (Iprivask™)

INTERVENTIONS:
Drug: Desirudin (Iprivask™) — Patients who are randomized to the desirudin (study) group will receive 15 mg of subcutaneous desirudin twice a day (at 0900 and 2100). These patients will also receive an injection of normal saline placebo at 1300 so that patients in both groups will receive three injections at the same time points.
  Arms: Desirudin (Iprivask™)
Drug: Heparin — The patients who are randomized to the Heparin (standard of care) group will receive subcutaneous injections of heparin three times a day (0900, 1300 and 2100).
  Arms: Heparin

SUMMARY:
A blood clot in the veins, also known as deep venous thrombosis (DVT), is one of the most common complications after surgery. This may result in death if a clot breaks off and travel to the lungs; this is referred to as pulmonary embolism (PE). After heart surgery the incidence of DVT ranges from 20-48% and following lung surgery the incidence is 19-26%. In order to decrease the likelihood of this complication, patients receive by injection a blood thinning medicine. Heparin is the usual medicine used for this purpose following heart and lung surgery. Recently there have been reports that other medicines may be more effective than heparin for this purpose. Also there have been reports that some patients develop antibodies to heparin. When this occurs, this may prevent the heparin from being effective and may even promote the formation of blood clots. Antibodies to heparin may be present more often following heart and lung surgery than other types of surgery. There is a new medicine called desirudin (Iprivask), which may be used instead of heparin to prevent blood clots following heart and lung surgery. Desirudin is currently approved by the FDA to prevent blood clots following hip surgery. The purpose of this study is to compare desirudin with heparin for the prevention of vein clots after heart and lung surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are scheduled for elective Cardiac or Thoracic Surgery.
* Age > 18 years of age.

Exclusion Criteria:

* Patients with a clinical suspicion or a documented history of DVT/PE
* Patients who may require anticoagulation during the post-op period. (i.e. Patients with a history of A-fib, scheduled for a MAZE procedure or placement of a mechanical valve, or those on Coumadin/IV heparin preoperatively)
* Patients who have a history of HIT or if there is a suspicion of the patient having HIT pre-operatively.
* Documented allergy to heparin, desirudin, or lepirudin
* Patients with a history of coagulation disorder
* Platelet count< 100 X109 /dl
* Active bleeding
* Serum Creatinine ≥ 1.5 mg/dl or CrCl ≤ 30 ml/min
* Patients with a baseline coagulopathy (INR > 1.5 or aPTT > 45 sec)
* Patients with liver disease
* Pregnancy
* Patients who require ventricular assist devices before or after surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2006-05; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael S Avidan, MBBCh, Principal Investigator — Washington University School of Medicine; Charles Hantler, MD, Study Director — Washington University School of Medicine; Bryan Meyers, MD, Study Chair — Washington University School of Medicine
Locations (1):
- Barnes-Jewish Hospital, St Louis, Missouri, United States

REFERENCES:
- [Derived] Graetz TJ, Tellor BR, Smith JR, Avidan MS. Desirudin: a review of the pharmacology and clinical application for the prevention of deep vein thrombosis. Expert Rev Cardiovasc Ther. 2011 Sep;9(9):1101-9. doi: 10.1586/erc.11.131. PMID 21932952
- [Derived] Avidan MS, Smith JR, Skrupky LP, Hill L, Jacobsohn E, Burnside B, Tymkew H, Eby C, Damiano R, Despotis GJ. The occurrence of antibodies to heparin-platelet factor 4 in cardiac and thoracic surgical patients receiving desirudin or heparin for postoperative venous thrombosis prophylaxis. Thromb Res. 2011 Dec;128(6):524-9. doi: 10.1016/j.thromres.2011.05.025. Epub 2011 Jul 26. PMID 21794899

RESULTS

PARTICIPANT FLOW:
Groups:
- Desirudin: Patients randomized to the desirudin group received desirudin 15mg via subcutaneous administration twice daily (0900 and 2100), with saline placebo given once daily at 1300.
- Heparin: Patients randomized to the heparin group received 5000 units of LDUH via subcutaneous administration three times a day (0900, 1300, and 2100).
Period: Overall Study
Arm/Group | Desirudin | Heparin
Started | 61 | 59
Completed | 61 | 59
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Desirudin | Heparin | Total
Number analyzed (Participants) | 61 | 59 | 120
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 38 | 39 | 77
  >=65 years | 23 | 20 | 43
Age, Continuous [Mean (Standard Deviation); unit: years] | 62 (11) | 61 (12) | 61 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 22 | 48
  Male | 35 | 37 | 72
Region of Enrollment [Number; unit: participants]
  United States | 61 | 59 | 120

OUTCOME MEASURES:

1. Primary Outcome: The Primary Outcome Measure Was the Number of Participants With New Heparin Platelet Factor 4 (HIT Positive) Antibodies in Each Group Within 30 Days Following Surgery.
Description: Blood samples were collected and tested in singlet for the presence of PF4/heparin antibodies. Samples were collected for each participant on PDD (Post-study Drug initiation Day) 2, PDD 7 or at hospital discharge, and at 30 days post surgery.
Time Frame: 30 days after surgery
Population: Intent-to-treat analysis was performed according to initial group assignment.
Measure: Number; unit: participants
Arm/Group | Desirudin | Heparin
Number analyzed (Participants) | 61 | 59
participants | 6 | 8
Statistical Analysis 1: Comparison: Desirudin vs Heparin; Published data show that the incidence of PF4/heparin EIA antibodies is approximately 40% (range, 20% to 60%) following cardiac surgery. We estimated that antibody formation would occur in approximately 20% of patients following thoracic surgery. Sixty patients in each group would provide 80% power to detect a decrease in the incidence of positive PF4/heparin EIA tests from 20% to 4% at an alpha level of <0.05; Test type: Superiority or Other; p < 0.05, Fisher Exact

2. Secondary Outcome: The Incidence of DVTs in Each Group.
Time Frame: 7 days after surgery
Population: 61 in Desirudin group and 59 in heparin group.
Measure: Count of Participants; unit: Participants
Arm/Group | Desirudin | Heparin
Number analyzed (Participants) | 61 | 59
Participants | 3 | 2
Statistical Analysis 1: Comparison: Desirudin vs Heparin; Test type: Superiority; p < 0.05, Fisher Exact

3. Secondary Outcome: The Incidence of Bleeding in Each Group.
Time Frame: Up to 30 days after surgery
Population: Intention to treat.
Measure: Count of Participants; unit: Participants
Arm/Group | Desirudin | Heparin
Number analyzed (Participants) | 61 | 59
Participants | 2 | 2
Statistical Analysis 1: Comparison: Desirudin vs Heparin; Test type: Superiority; p < 0.05, Fisher Exact

ADVERSE EVENTS:
Arm/Group | Desirudin | Heparin
Serious Adverse Events (participants affected / at risk) | 0/61 | 0/59
Other Adverse Events (participants affected / at risk) | 0/61 | 0/59

LIMITATIONS AND CAVEATS:
The study size was small and a surrogate end point was the primary outcome. The study was not powered to show statistical differences in clinical outcomes. Many patients received both desirudin and heparin during the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less